CLINICAL TRIAL: NCT01952080
Title: A 12-Week Pharmacokinetic, Safety, and Pharmacodynamic Study of Teduglutide in Pediatric Subjects Aged 1 Year Through 17 Years, With Short Bowel Syndrome Who Are Dependent on Parenteral Support
Brief Title: A Pharmacokinetic, Safety, and Pharmacodynamic Study of Teduglutide in Pediatric Subjects With Short Bowel Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED-C13-003
Record Dates: First submitted 2013-09-23; First posted 2013-09-27 (Estimated); Results first posted 2015-09-14 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Short Bowel Syndrome
Keywords: SBS; Pediatric SBS; Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome | interventions — teduglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- teduglutide (Experimental): Open label teduglutide, subcutaneously injected.
  Interventions: Drug: teduglutide
- Standard of Care (No Intervention)

INTERVENTIONS:
Drug: teduglutide — Open label intervention. Each subject will be assigned to receive 0.0125, 0.025, or 0.05 mg/kg/day for the duration of the study
  Arms: teduglutide

SUMMARY:
This will be an open label, 4-cohort study. Non-randomized subjects will receive teduglutide in each of the 3 active cohorts. An attempt will be made to enroll additional subjects into an observational cohort who will receive standard of care. Three doses of teduglutide are to be investigated for 12 weeks. All subjects will be screened prior to the start of treatment (SOT) to establish baseline characteristics including safety, eligibility and nutritional support parameters.

ELIGIBILITY:
Key Inclusion Criteria:

* Current history of SBS as a result of major intestinal resection, (eg, due to necrotizing enterocolitis, midgut volvulus, intestinal atresia, or gastroschisis) for at least 12 months prior to screening
* Short bowel syndrome that requires parenteral nutrition/intravenous (PN/IV) support
* Stable PN/IV support for at least 3 months prior to enrollment based upon the opinion of the investigator

Key Exclusion Criteria:

* Serial transverse enteroplasty or any other bowel lengthening procedure performed within the past 3 months
* Unstable absorption due to cystic fibrosis, untreated Hirschsprung's disease or known DNA abnormalities (ie, Familial Adenomatous Polyposis, Fanconi syndrome)
* Evidence of obstruction on upper gastrointestinal (GI) series done within 6 months prior to screening
* Major gastrointestinal surgical intervention within 3 months prior to screening (insertion of feeding tube or endoscopic procedure is allowed)

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2013-11-14 (Actual); Primary Completion 2015-01-09 (Actual); Study Completion 2015-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (19):
- United States (18):
  - Children´s Hospital of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - Mattel Children's Hospital UCLA, Department of Pediatric Gastroenterology, Los Angeles, California
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children at IU Health, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Mott Children's Hospital, University of Michigan, Ann Arbor, Michigan
  - Childrens Mercy Hospitals & Clinics Pediatric Gastroenterology, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Montefiore Medical Center, The Bronx, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Tennessee Health Science Center Le Bonheur Pediatric Specialists, Memphis, Tennessee
  - Monroe Carell, Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Texas Children's Hospital, Baylor College of Medicine, Houston, Texas
  - Seattle Childrens Hospital Gastroenterology and Hepatology, Seattle, Washington
  - University of Wisconsin School of Medicine and Public Health Surgery, Madison, Wisconsin
- Great Ormond Street Hospital for Children, London, United Kingdom

REFERENCES:
- [Derived] Fifi A, Raphael BP, Terreri B, Uddin S, Kaufman SS. Effects of Teduglutide on Diarrhea in Pediatric Patients with Short Bowel Syndrome-Associated Intestinal Failure. J Pediatr Gastroenterol Nutr. 2023 Nov 1;77(5):666-671. doi: 10.1097/MPG.0000000000003922. Epub 2023 Aug 22. PMID 37889619
- [Derived] Carter BA, Cohran VC, Cole CR, Corkins MR, Dimmitt RA, Duggan C, Hill S, Horslen S, Lim JD, Mercer DF, Merritt RJ, Nichol PF, Sigurdsson L, Teitelbaum DH, Thompson J, Vanderpool C, Vaughan JF, Li B, Youssef NN, Venick RS, Kocoshis SA. Outcomes from a 12-Week, Open-Label, Multicenter Clinical Trial of Teduglutide in Pediatric Short Bowel Syndrome. J Pediatr. 2017 Feb;181:102-111.e5. doi: 10.1016/j.jpeds.2016.10.027. Epub 2016 Nov 15. PMID 27855998

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: SOC- no teduglutide therapy
- Teduglutide 0.0125 mg/kg/Day: Cohort 1 - Teduglutide 0.0125 mg/kg/day
- Teduglutide 0.025 mg/kg/Day: Cohort 2 - Teduglutide 0.025 mg/kg/day
- Teduglutide 0.05 mg/kg/Day: Cohort 3 - Teduglutide 0.05 mg/kg/day
Period: Overall Study
Arm/Group | Standard of Care | Teduglutide 0.0125 mg/kg/Day | Teduglutide 0.025 mg/kg/Day | Teduglutide 0.05 mg/kg/Day
Started | 5 | 8 | 14 | 15
Treated | 5 | 8 | 14 | 15
Completed | 5 | 7 | 14 | 14
Not Completed | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Protocol Non-compliance | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Teduglutide 0.0125 mg/kg/Day | Teduglutide 0.025 mg/kg/Day | Teduglutide 0.05 mg/kg/Day | Total
Number analyzed (Participants) | 5 | 8 | 14 | 15 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.2 (0.45) | 5.1 (4.55) | 4.6 (3.43) | 4.5 (3.16) | 4.7 (3.5)
Age, Customized [Count of Participants; unit: Participants]
  1 to 3 years | 5 | 4 | 6 | 7 | 22
  4 to 12 years | 0 | 3 | 7 | 7 | 17
  13 to 17 years | 0 | 1 | 1 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 7 | 14
  Male | 3 | 6 | 11 | 8 | 28
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 8 | 14 | 12 | 39
  United Kingdom | 0 | 0 | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Parenteral Support [Parenteral Nutrition (PN)/Intravenous (IV)] Volume at Week 12
Description: Percent change in PN/IV from the Baseline Visit to Week 12 Visit.
Time Frame: Baseline, Week 12
Population: Percent change in PN/IV volume from baseline to Week 12 based on prescribed data - Intent-to-Treat Population (ITT), defined as all participants who were enrolled in the study.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Standard of Care | Teduglutide 0.0125 mg/kg/Day | Teduglutide 0.025 mg/kg/Day | Teduglutide 0.05 mg/kg/Day
Number analyzed (Participants) | 5 | 7 | 13 | 14
percent change | 7.38 (12.756) | -9.95 (21.625) | -37.34 (26.422) | -39.11 (40.792)

2. Primary Outcome: Percent Change in Parenteral Support (PN/IV) Volume at End of Treatment
Description: Percent change in PN/IV from the Baseline Visit to End of Treatment Visit.
Time Frame: Baseline, End of Treatment
Population: Percent change in PN/IV volume from baseline to End of Treatment based on prescribed data - Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Standard of Care | Teduglutide 0.0125 mg/kg/Day | Teduglutide 0.025 mg/kg/Day | Teduglutide 0.05 mg/kg/Day
Number analyzed (Participants) | 5 | 8 | 14 | 15
percent change | 7.38 (12.756) | -8.60 (20.380) | -35.61 (26.198) | -36.50 (40.585)

3. Primary Outcome: Percent Change in Parenteral Support (PN/IV) Volume at Week 16
Description: Percent change in PN/IV from the Baseline Visit to Week 16 Visit.
Time Frame: Baseline, Week 16
Population: Percent change in PN/IV volume from baseline to Week 16 based on prescribed data - Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Standard of Care | Teduglutide 0.0125 mg/kg/Day | Teduglutide 0.025 mg/kg/Day | Teduglutide 0.05 mg/kg/Day
Number analyzed (Participants) | 5 | 7 | 14 | 14
percent change | 3.92 (16.616) | -11.25 (21.196) | -33.85 (27.017) | -31.80 (39.264)

4. Primary Outcome: Absolute Change in Parenteral Support (PN/IV) Volume at Week 12
Description: Absolute change in PN/IV from the Baseline Visit to Week 12 Visit.
Time Frame: Baseline, Week 12
Population: Absolute change in PN/IV volume from baseline to Week 12 based on prescribed data - Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: Liters/week
Arm/Group | Standard of Care | Teduglutide 0.0125 mg/kg/Day | Teduglutide 0.025 mg/kg/Day | Teduglutide 0.05 mg/kg/Day
Number analyzed (Participants) | 5 | 7 | 13 | 14
Liters/week | 0.43 (0.746) | -0.50 (0.910) | -2.78 (1.985) | -2.57 (3.564)

5. Other Pre Specified Outcome: Percent Change in Enteral Support (EN) Volume From Baseline at Week 12
Description: Percent change in enteral support requirements at Week 12 (liters/week)
Time Frame: Baseline, Week 12
Population: Percent change of EN volume from baseline to Week 12 based on subject diary data - Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Standard of Care | Teduglutide 0.0125 mg/kg/Day | Teduglutide 0.025 mg/kg/Day | Teduglutide 0.05 mg/kg/Day
Number analyzed (Participants) | 3 | 4 | 12 | 8
percent change | 16.82 (14.921) | 23.50 (22.060) | 50.93 (61.416) | 57.96 (44.953)

6. Other Pre Specified Outcome: Percent Change in Enteral Support (EN) Volume From Baseline at Week 16
Description: Percent change in enteral support requirements at Week 16 (liters/week)
Time Frame: Baseline, Week 16
Population: Percent change of EN volume from baseline to Week 16 based on subject diary data - Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Standard of Care | Teduglutide 0.0125 mg/kg/Day | Teduglutide 0.025 mg/kg/Day | Teduglutide 0.05 mg/kg/Day
Number analyzed (Participants) | 4 | 1 | 11 | 9
percent change | 52.06 (66.194) | 60.30 | 43.98 (78.599) | 58.93 (63.927)

7. Other Pre Specified Outcome: Absolute Change in Enteral Support (EN) Volume From Baseline at Week 12
Description: Absolute change in enteral support requirements at Week 12 (liters/week)
Time Frame: Baseline, Week 12
Population: Absolute change of EN volume from baseline to Week 12 based on subject diary data - Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: Liters/week
Arm/Group | Standard of Care | Teduglutide 0.0125 mg/kg/Day | Teduglutide 0.025 mg/kg/Day | Teduglutide 0.05 mg/kg/Day
Number analyzed (Participants) | 4 | 7 | 12 | 12
Liters/week | 0.69 (0.715) | 2.67 (4.412) | 2.64 (3.220) | 0.97 (1.127)

8. Other Pre Specified Outcome: Absolute Change in Enteral Support (EN) Volume From Baseline at Week 16
Description: Absolute change in enteral support requirements at Week 16 (liters/week)
Time Frame: Baseline, Week 16
Population: Absolute change of EN volume from baseline to Week 16 based on subject diary data - Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: Liters/week
Arm/Group | Standard of Care | Teduglutide 0.0125 mg/kg/Day | Teduglutide 0.025 mg/kg/Day | Teduglutide 0.05 mg/kg/Day
Number analyzed (Participants) | 5 | 3 | 11 | 13
Liters/week | 0.84 (0.624) | 4.56 (5.384) | 2.47 (3.403) | 0.91 (0.968)

9. Primary Outcome: Absolute Change in Parenteral Support (PN/IV) Volume at End of Treatment
Description: Absolute change in PN/IV from the Baseline Visit to End of Treatment Visit.
Time Frame: Baseline, End of Treatment
Population: Absolute change in PN/IV volume from baseline to End of Treatment based on prescribed data - Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: Liters/week
Arm/Group | Standard of Care | Teduglutide 0.0125 mg/kg/Day | Teduglutide 0.025 mg/kg/Day | Teduglutide 0.05 mg/kg/Day
Number analyzed (Participants) | 5 | 8 | 14 | 15
Liters/week | 0.43 (0.746) | -0.43 (0.864) | -2.73 (1.916) | -2.4 (3.498)

10. Primary Outcome: Absolute Change in Parenteral Support (PN/IV) Volume at Week 16
Description: Absolute change in PN/IV from the Baseline Visit to Week 16 Visit.
Time Frame: Baseline, Week 16
Population: Absolute change in PN/IV volume from baseline to Week 16 based on prescribed data - Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: Liters/week
Arm/Group | Standard of Care | Teduglutide 0.0125 mg/kg/Day | Teduglutide 0.025 mg/kg/Day | Teduglutide 0.05 mg/kg/Day
Number analyzed (Participants) | 5 | 7 | 14 | 14
Liters/week | 0.17 (1.027) | -0.56 (0.885) | -2.56 (1.917) | -1.99 (3.092)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the first patient consent signed through last subject last visit for a duration of 421 days.
Description: This section reports "treatment-emergent" adverse events. Serious adverse events may be included in the 5% NSAE section.
Arm/Group | Standard of Care | Teduglutide 0.0125 mg/kg/Day | Teduglutide 0.025 mg/kg/Day | Teduglutide 0.05 mg/kg/Day
Serious Adverse Events (participants affected / at risk) | 3/5 | 3/8 | 6/14 | 8/15
Other Adverse Events (participants affected / at risk) | 5/5 | 8/8 | 14/14 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=5) | Teduglutide 0.0125 mg/kg/Day (N=8) | Teduglutide 0.025 mg/kg/Day (N=14) | Teduglutide 0.05 mg/kg/Day (N=15)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
Frequent Bowel Movement (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
Pyrexia (General disorders) | 2 (2) | 0 | 1 (1) | 3 (3)
Catheter related complication (General disorders) | 1 (1) | 0 | 2 (2) | 1 (1)
Fatigue (General disorders) | 0 | 0 | 0 | 1 (1)
Irritability (General disorders) | 0 | 0 (0) | 0 | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1 (1)
Central line infection (Infections and infestations) | 0 | 0 | 3 (5) | 1 (2)
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 1 (1) | 1 (1)
Adenovirus infection (Infections and infestations) | 0 | 1 (1) | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 1 (1) | 0 | 0
Catheter sepsis (Infections and infestations) | 0 | 0 | 0 | 1 (1)
Influenza (Infections and infestations) | 0 | 1 (1) | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1 (1) | 0
Fungaemia (Infections and infestations) | 1 (1) | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 (1) | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 (1) | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 (1)
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 1 (1) | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 0
Hypovolemic shock (Vascular disorders) | 0 | 0 | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Standard of Care (N=5) | Teduglutide 0.0125 mg/kg/Day (N=8) | Teduglutide 0.025 mg/kg/Day (N=14) | Teduglutide 0.05 mg/kg/Day (N=15)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 (2) | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 (2) | 0
Tachycardia (Cardiac disorders) | 1 (1) | 0 | 1 (1) | 1 (1)
Eyes sunken (Eye disorders) | 0 | 0 | 0 | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 | 0 | 5 (8) | 7 (29)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (5) | 4 (15)
Nausea (Gastrointestinal disorders) | 0 | 1 (3) | 2 (2) | 2 (8)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 | 1 (1) | 3 (6)
Faecal volume increased (Gastrointestinal disorders) | 0 | 1 (1) | 1 (1) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 | 1 (2) | 1 (1) | 1 (2)
Flatulence (Gastrointestinal disorders) | 0 | 2 (2) | 1 (1) | 0
Haematochezia (Gastrointestinal disorders) | 0 | 2 (2) | 1 (1) | 0
Constipation (Gastrointestinal disorders) | 1 (2) | 0 | 0 | 2 (2)
Painful defaecation (Gastrointestinal disorders) | 0 | 0 | 0 | 2 (2)
Retching (Gastrointestinal disorders) | 0 | 0 | 2 (2) | 0
Catheter related complication (General disorders) | 1 (1) | 3 (4) | 4 (4) | 2 (3)
Pyrexia (General disorders) | 2 (3) | 0 | 2 (2) | 7 (8)
Fatigue (General disorders) | 0 | 0 | 1 (1) | 4 (11)
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 3 (4)
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 2 (2) | 0
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (3) | 4 (6) | 4 (4)
Central line infection (Infections and infestations) | 0 | 0 | 3 (5) | 1 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1) | 0 | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 | 2 (2) | 0 | 1 (1)
Influenza (Infections and infestations) | 0 | 1 (1) | 1 (1) | 0
Overgrowth bacterial (Infections and infestations) | 0 | 2 (2) | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 1 (1) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 | 0 | 2 (2) | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0/0 | 0/1 | 0/1 | 1/1 (5) — Only 1 subject in each of the 3 dosing cohorts had a stoma and no standard of care subject had a stoma.
Feeding tube complication (Injury, poisoning and procedural complications) | 0 | 0 | 2 (2) | 0
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 1 (1)
Blood bicarbonate decreased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 3 (4)
Weight decreased (Investigations) | 0 | 1 (1) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 (1) | 1 (1)
Bacteria urine (Investigations) | 1 (1) | 0 | 0 | 2 (2)
Blood urine present (Investigations) | 0 | 0 | 0 | 2 (2)
Protein urine present (Investigations) | 0 | 0 | 0 | 2 (2)
Red blood cells urine positive (Investigations) | 0 | 0 | 0 | 2 (2)
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0 | 1 (1)
Headache (Nervous system disorders) | 0 | 1 (5) | 2 (2) | 2 (10)
Dizziness (Nervous system disorders) | 0 | 0 | 1 (1) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3) | 2 (3) | 4 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 (2) | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (3) | 2 (3)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 1 (1) | 1 (1)
Pallor (Vascular disorders) | 1 (1) | 0 | 0 (0) | 1 (1)
Fungaemia (Infections and infestations) | 1 (2) | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0 | 0
White blood cell count increased (Investigations) | 1 (1) | 0 | 0 | 0
Urine leukocyte esterase positive (Investigations) | 1 (1) | 0 | 0 | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 | 0 | 1 (1)
Gastrointestinal bacterial infection (Infections and infestations) | 1 (1) | 0 | 0 | 0
Irritability (General disorders) | 1 (1) | 0 | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No